CLINICAL TRIAL: NCT01146886
Title: A Randomised, Double-blind, Placebo-controlled Trial to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of 10 mg to 1200 mg of BI 135585 XX Administered as a Solution to Healthy Male Volunteers (Trial Part 1), Followed by an Open, Randomised, Single-dose, Intra-individual Bioavailability Comparison of 200 mg BI 135585 XX as Tablet and as Solution (Trial Part 2)
Brief Title: Trial to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Oral Doses of BI135585 XX Administered as Tablet and as Solution in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1283.1; 2010-018856-28 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-06-14; First posted 2010-06-22 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 6-(2-hydroxy-2-methylpropyl)-3-(1-(4-(1-methyl-2-oxo-1,2-dihydropyridin-4-yl)phenyl)ethyl)-6-phenyl-1,3-oxazinan-2-one

ARMS (2):
- BI 135585 (Experimental): 1 single dose per subject as oral solution in Part 1, or 3 single doses per subject as oral solution and 2 different tablet formulations in Part 2
  Interventions: Drug: BI 135585
- Placebo to BI 135585 (Placebo Comparator): 1 single dose per subject as oral solution in Part 1
  Interventions: Drug: Placebo to BI 135585

INTERVENTIONS:
Drug: Placebo to BI 135585 — Part 1 - oral doses given to approximately 9 parallel groups of 8 subjects (6 on active and 2 on on placebo) on Day 1
  Arms: Placebo to BI 135585
Drug: BI 135585 — Part 1 - oral doses given to approximately 9 parallel groups of 8 subjects (6 on active and 2 on placebo) on Day 1; Part 2 - oral doses given to 12 subjects on Day 1
  Arms: BI 135585

SUMMARY:
The purpose of the study is to investigate the safety, tolerability, pharmacokinetics incl. dose proportionality, and pharmacodynamics of BI 135585 XX (Part 1), as well as the relative bioavailability of two different immediate release tablet formulations versus oral solution (Part 2)

ELIGIBILITY:
Inclusion criteria:

- healthy male volunteers

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Physical examination (occurrence of findings) | up to 14 days post treatment
Change from baseline in Vital signs (blood pressure [BP], pulse rate [PR], respiratory rate [RR]) | up to 14 days post treatment
Change from baseline in 12-lead ECG with special attention to QTc prolongation | up to 14 days post treatment
Cardiopulmonary monitoring resulting in clinically relevant findings | up to 14 days post treatment
Change from baseline in Clinical laboratory parameters including hormones of the HPA axis and thyroid gland | up to 14 days post treatment
Number of patients with Adverse events (AE) | up to 14 days post treatment
Assessment of tolerability by the investigator | up to 14 days post treatment

SECONDARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 72 hours post treatment
(5α-THF + 5β-THF)/THE ratio as an indicator of 11β-HSD1 inhibition | up to 24h
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 72 hours post treatment
Cmax (maximum measured concentration of the analyte in plasma) | up to 72 hours post treatment
tmax (time from dosing to maximum measured concentration) | up to 72 hours post treatment
%AUCtz-∞ (percentage of the AUC0-∞ that was obtained by extrapolation) | up to 72 hours post treatment
λz (terminal rate constant in plasma) | up to 72 hours post treatment
t1/2 (terminal half-life of the analyte in plasma) | up to 72 hours post treatment
MRToral (mean residence time of the analyte in the body after oral administration) | up to 72 hours post treatment
CL/F (total/apparent clearance of the analyte in plasma after extravascular administration) | up to 72 hours post treatment
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 72 hours post treatment
Aet1-t2 (amount of analyte eliminated in urine from timepoint t1 to timepoint t2) SRD part only | up to 72 hours post treatment
fet1-t2 (fraction of analyte eliminated in urine from timepoint t1 to timepoint t2) SRD part only | up to 72 hours post treatment
CLR,t1-t2 (renal clearance of the analyte from timepoint t1 to timepoint t2) SRD part only[ | up to 72 hours post treatment
UFF/UFE ratio as an indicator of 11β-HSD2 inhibition | up to 24h
Total urinary corticosteroids (5α-THF + 5β-THF + THE + UFF + UFE) as an indicator of the activation of the HPA axis | up to 24h

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1283.1.1 Boehringer Ingelheim Investigational Site, Biberach, Germany